CLINICAL TRIAL: NCT02182778
Title: Randomized Phase III Trial Comparing Gemcitabine/Cisplatin/S-1 With Gemcitabine/Cisplatin for Unresectable Biliary Tract Cancer
Brief Title: GEM/Cisplatin/S-1 vs GEM/Cisplatin for Biliary Tract Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1401; UMIN 000014371 (Registry Identifier: UMIN)
Record Dates: First submitted 2014-06-28; First posted 2014-07-08 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2018-04

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine/Cisplatin group (Experimental): Gemcitabine and cisplatin are infused on day1, 8. The cycle is repeated every 3 weeks.
  Interventions: Drug: Gemcitabine/Cisplatin /S-1
- Gemcitabine/Cisplatin /S-1 group (Experimental): S-1 is given daily for 7 consecutive days and gemcitabine and cisplatin are infused on day1. The cycle is repeated every 2 weeks.
  Interventions: Drug: Gemcitabine/Cisplatin

INTERVENTIONS:
Drug: Gemcitabine/Cisplatin — Gemcitabine and cisplatin are infused on day1, 8. The cycle is repeated every 3 weeks.
  Other Names: Gemcitabine;gemzer, Cisplatin;Cispulan
  Arms: Gemcitabine/Cisplatin /S-1 group
Drug: Gemcitabine/Cisplatin /S-1 — S-1 is given daily for 7 consecutive days and gemcitabine and cisplatin are infused on day1. The cycle is repeated every 2 weeks.
  Other Names: Gemcitabine;gemzer, Cisplatin;Cispulan S-1;TS-1,
  Arms: Gemcitabine/Cisplatin group

SUMMARY:
To validate the superiority of Gemcitabine/Cisplatin/S-1 over Gemcitabine/Cisplatin for unresectable biliary tract cancer.

DETAILED DESCRIPTION:
Gemcitabine/cisplatin combination therapy (GC) has been the standard palliative chemotherapy for patients with advanced biliary tract cancer (BTC). Investigators have evaluated the efficacy and safety of gemcitabine/cisplatin/S-1 combination therapy (GCS) for patients with advanced BTC and observed the promising efficacy. In this randomized phase Ⅲ study, investigators aimed to compare GCS with GC in patients with advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cytologically or histologically proved biliary tract cancer
2. age >=20 years
3. Performance Status (PS) 0-2
4. No prior history of chemotherapy or radiotherapy.
5. Adequate bone marrow function (neutrophil count >=1,500/mm3, and platelet count >=100,000/mm3), liver function (total bilirubin >=3 mg/dL and AST/ALT >=150 IU/L), and renal function (creatinine clearance >=45 mL/min)
6. Adequate oral intake
7. Provided written informed consent -

Exclusion Criteria:

1. Patients with interstitial pneumonia or pulmonary fibrosis
2. Patients with uncontrollable diabetes mellitus, liver disease, angina pectoris or a new onset of myocardial infarction within 3 months
3. Patients with severe active infection
4. Patients with moderate or marked pleural effusion or ascites necessitating drainage
5. Patients with a history of severe drug allergy
6. Patients with other serious comorbid disease
7. Patients who are pregnant or lactating, or have an intention to get pregnant
8. Patients with mental disease
9. Patients who are judged inappropriate for the entry into the study by the principle doctor

   -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2016-02-04 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | Probability of 1-year survival (%)
  The primary endpoint is designated to evaluate overall survival rate at 12-month.

SECONDARY OUTCOMES:
Response rate | Every 3 months, up to 24 months
  The investigators will conduct CT test every 3 months in order to measure the tumor size of each patient and evaluate the best tumor response according to RECIST criteria.
Progression free survival | Every 3 months, up to 24 months
  In oredr to research the progression survival, the investigators will check the presence of progression disease for each patient every three months.
Number of Participants with Adverse Events as a Measure of Safety | 24 months
  The investigators will examine the frequency and the degree of each side effect that will appear to the patient at each course of chemotherapy .

CONTACTS AND LOCATIONS:
Overall Officials: Masashi Kanai, Study Director — Kyoto University
Locations (1):
- Kyoto University Hospital, Kyoto, Japan

REFERENCES:
- [Derived] Ioka T, Kanai M, Kobayashi S, Sakai D, Eguchi H, Baba H, Seo S, Taketomi A, Takayama T, Yamaue H, Takahashi M, Sho M, Kamei K, Fujimoto J, Toyoda M, Shimizu J, Goto T, Shindo Y, Yoshimura K, Hatano E, Nagano H; Kansai Hepatobiliary Oncology Group (KHBO). Randomized phase III study of gemcitabine, cisplatin plus S-1 versus gemcitabine, cisplatin for advanced biliary tract cancer (KHBO1401- MITSUBA). J Hepatobiliary Pancreat Sci. 2023 Jan;30(1):102-110. doi: 10.1002/jhbp.1219. Epub 2022 Aug 9. PMID 35900311
- [Derived] Kanai M, Hatano E, Kobayashi S, Fujiwara Y, Marubashi S, Miyamoto A, Shiomi H, Kubo S, Ikuta S, Yanagimoto H, Terajima H, Ikoma H, Sakai D, Kodama Y, Seo S, Morita S, Ajiki T, Nagano H, Ioka T. A multi-institution phase II study of gemcitabine/cisplatin/S-1 (GCS) combination chemotherapy for patients with advanced biliary tract cancer (KHBO 1002). Cancer Chemother Pharmacol. 2015 Feb;75(2):293-300. doi: 10.1007/s00280-014-2648-9. Epub 2014 Dec 5. PMID 25477010